CLINICAL TRIAL: NCT01299012
Title: Liraglutide as Additional Treatment in Patients With Type 1 Diabetes Mellitus, a Retrospective Chart Review
Brief Title: Liraglutide as Additional Treatment in Patients With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Paresh Dandona, MD, Kaleida Health
Other Study IDs: 1954
Record Dates: First submitted 2011-02-01; First posted 2011-02-18 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Liraglutide — Liraglutide s/c 0.6mg once daily.
  Other Names: Victoza

SUMMARY:
Evaluating the use of Liraglutide in patients with Type 1 Diabetes.

DETAILED DESCRIPTION:
This investigation will be a retrospective chart review of in type 1 diabetics who have been treated with liraglutide. The study will be conducted at Diabetes-Endocrinology Center of WNY at Millard Fillmore Hospital, affiliated to the State University of New York at Buffalo.

Study Population: 40 patients with type 1 diabetes on treatment with either continuous subcutaneous insulin infusion (CSII; also known as insulin pump) or multiple (four or more) injections of insulin per day on continuous glucose monitoring system (CGMS) will be included in the study. These patients with type 1 diabetes have been treated with liraglutide in addition to insulin. The investigators would retrospectively review their charts to evaluate decreases in fasting, postprandial and the overall mean glucose concentrations.

The investigators will compare the mean fasting, the mean weekly glucose and the standard deviation of weekly blood glucose concentrations as recorded by continuous glucose monitoring prior to and following one week and 12 weeks of treatment with liraglutide daily. In addition, the investigators will compare the time spent at glucose concentrations >150 and 200mg/dl and <70 and <40 mg/dl. HbA1c levels before and after 12 weeks of treatment with liraglutide daily will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus

Exclusion Criteria:

* Type 2 Diabetes Mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 Diabetes Mellitus
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Improved Blood Glucose comtrol in Type 1 Diabetes Patients with Liraglutide | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, Principal Investigator — University at Buffalo